CLINICAL TRIAL: NCT00493506
Title: The Effects of ProAlgaZyme Novel Algae Infusion Alone or in Combination With HAART on Markers of Immune Status, Dyslipidemia, Inflammation and Oxidative Stress in HIV or HIV/HBV Patients
Brief Title: ProAlgaZyme Novel Algae Infusion: Applications in Immunodeficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Enhancement Products, Inc. (Industry)
Collaborators: University of Yaounde (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-0002-01; 087/2006
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2007-06-28 (Estimated); Status verified 2007-06

CONDITIONS: HIV Infections; Hepatitis B; Dyslipidemia
Keywords: ProAlgaZyme; HIV; HAART; hsCRP; Oxidative stress; CD4+ lymphocytes; Algae; HAART adverse effects; HBV
MeSH Terms: conditions — HIV Infections; Hepatitis B; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ProAlgaZyme

SUMMARY:
The purpose of this study is to determine the safety and effects in HIV patients of supplementation (4-20 fl. oz. daily) with ProAlgaZyme, a novel fermentation product of a freshwater algae ecosystem, on markers of immune status, dyslipidemia, inflammation and oxidative stress alone or in combination with HAART (highly-active antiretroviral therapy).

DETAILED DESCRIPTION:
HIV infection and interventions such as HAART (highly-active antiretroviral therapy) are associated with dyslipidemia and increased markers of inflammatory and oxidative stress. These effects can hasten the progression towards AIDS and present serious cardiovascular complications. Therapeutic agents that can provide immune support with minimal side effects and/or reduce the adverse effects of HAART are in high demand worldwide. Such agents may help HIV patients to live a better quality of life, and may potentially improve the compliance with traditional therapies including HAART. This study is a single-center open-label design to evaluate the safety of ProAlgaZyme novel algae infusion and its effects in varying dosages on markers of immune status, dyslipidemia, inflammation and oxidative stress in patients with HIV or HIV/HBV co-infection, who may also be taking HAART.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as HIV +ve or HIV/HBV +ve
* Either/or:

  * had not taken antiretroviral drugs before (pre-HAART patients)
  * were treated with triple drug therapy for at least 3-6 months

Exclusion Criteria:

* Obese
* Taking any cholesterol-lowering medications 30 days prior to the start of enrollment and during the course of the study.
* Enrolled in another clinical study in the past 6 months.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2006-05; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
CD4+ T-lymphocytes | 12 weeks
HIV Viral Load | 12 weeks
hsCRP (C-reactive protein) | 12 weeks
Total cholesterol | 12 weeks
Liver enzymes (ALT, ALP, GGT) | 12 weeks
MDA (malonaldehyde) and thiol proteins | 12 weeks

SECONDARY OUTCOMES:
RBC and WBC counts | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Julius Oben, Ph.D., Principal Investigator — Laboratory of Nutrition and Nutritional Biochemistry (LNNB), Department of Biochemistry, University of Yaounde I, Yaounde, Cameroon
Locations (1):
- Laboratory of Nutrition and Nutritional Biochemistry (LNNB), Department of Biochemistry, University of Yaounde I, Yaoundé, Cameroon